CLINICAL TRIAL: NCT04500808
Title: A Double-blind, Randomized, Placebo-controlled, Multiple-dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Macitentan and an Open-label, Randomized, Crossover, Single-dose Study to Evaluate the Effect of Food on Macitentan Pharmacokinetics, in Healthy Japanese Adult Male Participants
Brief Title: A Study of Macitentan, in Healthy Japanese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CR108788; 67896062PAH1005 (Other: Janssen Pharmaceutical K.K., Japan)
Record Dates: First submitted 2020-07-17; First posted 2020-08-05 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1: Double Blind Phase (Experimental): Participants will receive macitentan or matching placebo from Day 1 up to Day 13 under fed conditions and will be up-titrated starting with 2 once daily (QD) dosing of Dose 1 from Days 1 to 2 followed by 3 qd doses of Dose 2 of macitentan from Days 3 to 5, followed by qd doses of Dose 3 macitentan from Days 6 to 13.
  Interventions: Drug: Macitentan Dose 1; Drug: Macitentan Dose 2; Drug: Macitentan Dose 3; Drug: Placebo
- Part 2: Open Label Phase: Treatment Sequence AB (Experimental): Participants will receive Dose 3 of macitentan under fasted conditions (Treatment A) in period 1 followed by Dose 3 of macitentan under fed condition (Treatment B) in period 2 on Day 1 with a washout phase of at least 14 days between the two treatment periods.
  Interventions: Drug: Macitentan Dose 3
- Part 2: Open Label Phase: Treatment Sequence BA (Experimental): Participants will receive Treatment B in period 1 followed by Treatment A in period 2 on Day 1 with a washout phase of at least 14 days between the two treatment periods.
  Interventions: Drug: Macitentan Dose 3

INTERVENTIONS:
Drug: Macitentan Dose 1 — Participants will receive Dose 1 of macitentan tablet in Part 1.
  Other Names: JNJ-67896062
  Arms: Part 1: Double Blind Phase
Drug: Macitentan Dose 2 — Participants will receive Dose 2 of macitentan tablet in Part 1.
  Other Names: JNJ-67896062
  Arms: Part 1: Double Blind Phase
Drug: Macitentan Dose 3 — Participants will receive Dose 2 of macitentan tablet in Part 1 and 2.
  Other Names: JNJ-67896062
Drug: Placebo — Participants will receive matching placebo from Day 1 up to Day 13.
  Arms: Part 1: Double Blind Phase

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability after multiple-dose administrations of macitentan with titration regimen starting from Dose 1 once daily (qd) up to Dose 2 qd in Japanese healthy adult male participants (Part 1) and to evaluate the effect of food on pharmacokinetics of macitentan and its active metabolite (ACT-132577) in Japanese healthy adult male participants with macitentan Dose 3 tablet (Part 2).

ELIGIBILITY:
Inclusion Criteria:

* Be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel, hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities or deviations from normal to be not clinically significant. This determination must be recorded in the participant's source documents and initialed by the investigator
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic
* A participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person. Male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak. Recommended highly effective methods of contraception in this study for female partners of male participants to use in addition to the male participant wearing a condom during include: oral hormonal contraception, intrauterine device, intrauterine hormone-releasing system and bilateral tubal occlusion
* A participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum 90 Days after receiving the last dose of study intervention
* Nonsmoker or smoker habitually smokes no more than 10 cigarettes or equivalent of e-cigarettes, or 2 cigars, or 2 pipes of tobacco per day for at least 6 months before first study drug administration

Exclusion Criteria:

* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency (creatinine clearance below 80 (milliliter per minute) mL/min calculated using Cockcroft-Gault equation), thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening or at admission to the study site as deemed appropriate by the investigator
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin or malignancy, which is considered cured with minimal risk of recurrence)
* Known allergies, hypersensitivity, or intolerance to macitentan or its excipients
* Known allergy to heparin or history of heparin-induced thrombocytopenia

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) | Up to Day 29
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Part 1: Number of Participants with Adverse Event of Special Interests (AESIs) | Up to Day 29
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. The following are the AEs of special interest in this study: Hypotension: symptomatic hypotension or potentially clinically meaningful decrease in blood pressure, Edema/fluid retention: clinically relevant signs and symptoms of edema and/or fluid retention, Hemoglobin decrease/anemia: events of hemoglobin decrease from baseline of greater than (>) 20 gram per liter (g/L), Liver events: liver aminotransferase abnormalities.
Part 1: Number of Participants with Serious Adverse Events (SAEs) | Up to Day 29
  A SAE is any AE that results in: death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is a suspected transmission of any infectious agent via a medicinal product, is medically important.
Part 1: Number of Participants with Clinical Laboratory Abnormalities | Up to Day 29
  Number of participants with clinical laboratory abnormalities (serum chemistry, hematology, blood coagulation) will be reported
Part 1: Number of Participants with Abnormalities in ECG Variables | Up to Day 29
  Number of Participants with abnormalities in ECG variables such as: PR, QRS, QT, RR, and QT corrected Fridericia's formulae (QTcF) will be reported.
Part 1: Change from Baseline in Weight | Baseline, up to Day 29
  Change from baseline in body weight in kilograms as a part of physical examination will be reported.
Part 1: Change from Baseline in Height | Baseline, up to Day 29
  Change from baseline in height in centimeters as a part of physical examination will be reported.
Part 2: Plasma Concentration of Macitentan and its Active Metabolite (ACT-132577) | Predose, 3, 5, 7, 8, 9, 10, 12, 16, 24, 48, 72, 120, 168, and 240 hours post dose
  Plasma concentration of macitentan and its active metabolite (ACT-132577) will be reported.

SECONDARY OUTCOMES:
Part 1: Plasma Concentration of Macitentan and its Active Metabolite (ACT-132577) | Day 5 and Day 13 (predose,1, 3, 5, 7, 8, 9, 10, 12, and 16 hours postdose)
  Plasma concentration of macitentan and its active metabolite (ACT-132577) will be reported.
Part 1: Plasma Endothelin-1 (ET-1) Concentrations | Up to Day 29
  Plasma ET-1 concentrations for macitentan and ACT-132577 will be reported.
Part 2: Number of Participants with Adverse Events (AEs) | Up to Day 12
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Part 2: Number of Participants with Adverse Event of Special Interests (AESIs) | Up to Day 12
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal product. An AE does not necessarily have a causal relationship with the intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product. The following are the AEs of special interest in this study: Hypotension: symptomatic hypotension or potentially clinically meaningful decrease in blood pressure, Edema/fluid retention: clinically relevant signs and symptoms of edema and/or fluid retention, Hemoglobin decrease/anemia: events of hemoglobin decrease from baseline of greater than (>) 20 gram per liter (g/L), Liver events: liver aminotransferase abnormalities.
Part 2: Number of Participants with Serious Adverse Events (SAEs) | Up to Day 12
  A SAE is any AE that results in: death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect and is a suspected transmission of any infectious agent via a medicinal product, is medically important.
Part 2: Number of Participants with Clinical Laboratory Abnormalities | Up to Day 12
  Number of participants with clinical laboratory abnormalities (serum chemistry, hematology, blood coagulation, and urine samples) will be reported
Part 2: Number of Participants with Abnormalities in ECG Variables | Up to Day 12
  Number of Participants with abnormalities in ECG variables such as: PR, QRS, QT, RR, and QT corrected Fridericia's formulae (QTcF) will be reported.
Part 2: Change from Baseline in Weight | Baseline, Up to Day 12
  Change from baseline in body weight in kilograms as a part of physical examination will be reported.
Part 2: Change from Baseline in Height | Baseline, Up to Day 12
  Change from baseline in height in centimeters as a part of physical examination will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Sumida Hospital, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency